CLINICAL TRIAL: NCT04627142
Title: A Phase 1 Open-label Dose Escalation Trial of BI 1701963 in Combination With Irinotecan in KRAS Mutation Positive Patients With Unresectable Locally Advanced or Metastatic Colorectal Cancer
Brief Title: A Study to Test Different Doses of BI 1701963 in Combination With Irinotecan in People With Advanced Bowel Cancer With Kirsten Rat Sarcoma Viral Oncogene Homologue (KRAS) Mutation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1432-0008
Record Dates: First submitted 2020-11-10; First posted 2020-11-13 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Intervention Model Description: Trial consists of three parts: Monotherapy safety run-in part (Part A), combination dose escalation part (Part B), combination therapy expansion part (Part C). A randomization will be included for the expansion therapy part (Part C) because the same patient population will be recruited to two different dose levels at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expansion dose 1 (Experimental): Part C: Combination therapy expansion part
  Interventions: Drug: BI 1701963; Drug: Camptosar®
- Expansion dose 2 (Experimental): Part C: Combination therapy expansion part
  Interventions: Drug: BI 1701963; Drug: Camptosar®

INTERVENTIONS:
Drug: BI 1701963 — Tablet
Drug: Camptosar® — Solution for infusion

SUMMARY:
This study is open to adults with advanced bowel cancer (colorectal cancer) with a KRAS mutation. This is a study in people for whom previous treatment was not successful and surgery is not a treatment option.

The purpose of this study is to find the highest dose of BI 1701963 that people with bowel cancer can tolerate when taken together with a medicine called irinotecan. The study also tests whether BI 1701963 in combination with irinotecan is able to make tumours shrink. BI 1701963 may help to turn off KRAS. Activating KRAS mutations make tumours grow. Irinotecan is a medicine to treat bowel cancer.

Participants can stay in the study as long as they benefit from treatment and can tolerate it.

During this time, participants take BI 1701963 as tablet once a day and get irinotecan as infusion every two weeks. The doctors regularly monitor the size of the tumour. The doctors also collect information on any health problems of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a confirmed activating KRAS mutation in CRC tumour tissue by local test. Activating mutations include but are not limited to: KRAS mutations in exon 2 (G12, G13), exon 3 (A59, Q61) and exon 4 (K117, A146)
* Patients must have a histological or cytological diagnosis of CRC
* Patients must have received at least first-line chemotherapy (oxaliplatin/ 5-Fluorouracil (5-FU)/ capecitabine et al treatment failure) for unresectable locally advanced or metastatic CRC
* Must have at least one target lesion that can be accurately measured per RECIST version 1.1
* Must have Eastern Cooperative Oncology Group score of 0 or 1
* Must show adequate organ function defined as all of the following:

  1. Absolute neutrophil count (ANC) ≥1.5 x 109/L; haemoglobin ≥9.0 g/dL; platelets ≥100 x 109/L without the use of hematopoietic growth factors within 4 weeks of start of Trial medication.
  2. Total bilirubin ≤1.5 x Upper Limited of Normal (ULN), or ≤4 x ULN for patients who are known to have Gilbert's syndrome
  3. Creatinine ≤1.5 x ULN. If creatinine is >1.5 x ULN, patient is eligible if concurrent glomerular filtration rate (GFR) ≥30 mL/min (measured or calculated by CKD-EPI formula)
  4. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤3 x ULN if no demonstrable liver metastases, or otherwise ≤5 x ULN
* For patients participating in the combination dose escalation and expansion parts (Part B and C), must be eligible to receive treatment with irinotecan in accordance with the local label including Summary of Product Characteristics (SmPC), U.S. PI or Chinese Label
* Must be at least 18 years of age at screening
* Must have recovered from any previous therapy related toxicity to CTCAE grade ≤1 before the first dose (except for alopecia; stable sensory neuropathy must be CTCAE grade ≤2)
* Signed and dated written informed consent in accordance with good clinical practice and local legislation prior to admission to the trial
* further inclusion criteria apply

Exclusion Criteria:

* Previous anticancer chemotherapy, anticancer immunotherapy, and/or other anticancer biologic therapy within 3 weeks of the first administration of trial drug. Previous anticancer hormonal therapy within 2 weeks of first administration of trial drug
* Previous treatment with a RAS, Mitogen-activated protein kinase (MAPK) or Son of Sevenless 1 (SOS1) targeting agent
* For patients participating in the combination dose escalation and expansion parts (Part B and C only): Previous treatment with irinotecan
* Radiotherapy within 4 weeks except as follows

  * Palliative radiotherapy to regions other than the chest is allowed up to 2 weeks prior to start of treatment
  * Single dose palliative radiotherapy for symptomatic metastasis within 2 weeks prior to start of treatment may be allowed but must be discussed with the sponsor
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to start of treatment or planned during the projected course of the trial, e.g. hip replacement
* Previous treatment with any investigational agent(s) or targeted treatment within 28 days prior to start of treatment
* Known history of hypersensitivity to any of the excipients of BI 1701963 tablets
* History or presence of cardiovascular abnormalities such as uncontrolled Hypertension, congestive heart failure New York Heart Association (NYHA) classification of ≥3, unstable angina or poorly controlled arrhythmia which are considered as clinically relevant by the investigator; Myocardial infarction within 6 months prior to start of treatment
* Left ventricular ejection fraction (LVEF) <50%
* Congenital long QT prolongation syndrome or mean resting corrected QT interval (QTcF) >470 msec
* further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) based on the number of dose limiting toxicities (DLTs) in the MTD evaluation period | 28 days
  Combination dose escalation part (Part B)
Number of patients experiencing DLTs in the MTD evaluation period | 28 days
  Combination dose escalation part (Part B)
Objective Response (OR) according to RECIST version 1.1 | 28 days per treatment cycle.
  Combination therapy expansion part (Part C)

SECONDARY OUTCOMES:
Number of patients with DLTs in the first treatment cycle | 28 days
  Monotherapy safety run-in part (Part A)
Maximum measured concentration of BI 1701963 in plasma (Cmax) | 28 days per treatment cycle.
  Monotherapy safety run-in part (Part A)
Area under the concentration time curve of BI 1701963 in plasma over the time interval from 0 to the last quantifiable plasma concentration (AUC0-tz) | 28 days per treatment cycle.
  Monotherapy safety run-in part (Part A)
Area under the concentration-time curve of BI 1701963 in plasma over the dosing interval τ at steady state (AUCτ(,ss)) | 28 days per treatment cycle.
  Monotherapy safety run-in and combination dose escalation part (Part A+B)
Maximum measured concentration of BI 1701963 in plasma at steady state over a uniform dosing interval tau (Cmax,ss) | 28 days per treatment cycle.
  Monotherapy safety run-in and combination dose escalation part (Part A+B)
Duration of objective response (DOR) | 28 days per treatment cycle.
  Combination therapy expansion part (Part C)
Tumour shrinkage (in millimetres) | 28 days per treatment cycle.
  Combination therapy expansion part (Part C)
Progression-free survival (PFS) | Up to 6 months.
  Combination therapy expansion part (Part C)
Number of patients experiencing grade ≥3 treatment-related AEs during the entire treatment period | 28 days per treatment cycle.
  Combination therapy expansion part (Part C)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Tongji University China, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/